CLINICAL TRIAL: NCT03464292
Title: Spinal and Supra-Spinal Pain Mechanisms in Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201800479; OCR17639 (Other: University of Florida)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Vehicle Patch: Control patch will be the same topical solution but will not contain capsaicin. The patch will applied to the hand for 30 - 60 min. Patients will be instructed to not touch or wash their hands during the course of the study to minimize spreading of the patch to other areas of the body. Subsequently, the patch will be immediately removed.
  Interventions: Other: Vehicle Patch
- Capsaicin Patch 8% or 0.1% Capsaicin Cream: 8% capsaicin topical patch or 0.1% capsaicin cream. The patch will applied to the hand for 30 - 60 min. The cream will be applied similarly on a 3 cm2 area of the arm. Patients will be instructed to not touch or wash their hands during the course of the study to minimize spreading of the patch to other areas of the body. Subsequently, the patch will be immediately removed.
  Interventions: Drug: Capsaicin Patch 8% or 0.1% Capsaicin Cream

INTERVENTIONS:
Drug: Capsaicin Patch 8% or 0.1% Capsaicin Cream — 0.1 ml of 8% capsaicin topical patch or 0.1% capsaicin cream
  Other Names: Qutenza; Capsaicin No-Fuss
  Groups: Capsaicin Patch 8% or 0.1% Capsaicin Cream
Other: Vehicle Patch — Control patch will be the same topical solution but will not contain capsaicin.
  Groups: Vehicle Patch

SUMMARY:
Fibromyalgia (FM) patients have increased windup (WU). However, WU of FM patients is only quantitatively but not qualitatively different from healthy controls (HC). Thus WU abnormalities of FM patients could be the result of supra-spinal and not the result of spinal pain mechanisms. The study team will test this hypothesis by sensitizing FM patients with topical capsaicin.

DETAILED DESCRIPTION:
The study team hypothesizes that at baseline the slopes of sensitivity adjusted WU of FM patients are not statistically different from HC. However, after capsaicin application, the slopes of sensitivity adjusted WU will be significantly different from baseline and greater than those of HC, suggesting central sensitization. This would imply that FM patients are sensitive to heat pain but not sensitized.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with fibromyalgia will have pain of duration > 6 months and meeting the 1990 Research Diagnostic Criteria for FM (ACR).
* healthy, pain-free age matched controls without chronic pain

Exclusion Criteria:

* Allergy to red chili peppers;
* Pregnant;
* Significant hearing loss;
* Presence of chronic disease (e.g. cancer, cardiovascular disease, liver disease, kidney disease, diabetes, etc.).
* FM patients must be willing to discontinue or hold their FM related medications for at least 5 half-lives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents living in or near Gainesville, FL
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Progression of Temporal Summation of Second Pain | 2 hr
  A Peltier device (Pathway, Medoc) will be used to tap the skin surface with a 3 cm x 3 cm probe. The Peltier device will be used to provide very brief, repetitive, thermal stimuli (for approx. 1s) to the skin using computer controlled temperatures. Heat stimuli at intervals of 2.5 sec produce sensations of increasing pain (temporal summation), depending on the number of stimuli presented. The late sensations of warmth are delayed in onset by approximately 1.5 sec after the probe touches the skin, because the sensation depends upon stimulation of slowly conducting unmyelinated peripheral afferents.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No